CLINICAL TRIAL: NCT05906238
Title: Development, Implementation and Evaluation of Interventions to Remediate the Threatening Effects of Obesity Stereotyes
Brief Title: Interventions to Remedy the Negative Effects of Obesity Stigma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STEREOBES
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Stigma, Weight
Keywords: Obesity; Therapeutic patient education; Stigmatization
MeSH Terms: conditions — Obesity; Weight Prejudice; Stereotyping

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STEREOBES (Experimental): This arm will follow a program developed specifically for this project. It will include specific workshops on obesity stigma issues which are not part of the standard program.
  Interventions: Behavioral: STEREOBES Workshops
- CONTROL (Active Comparator): This arm will follow the standard therapeutic patient education program proposed by "La Vie La Santé".
  Interventions: Behavioral: Un Poids en moins

INTERVENTIONS:
Behavioral: STEREOBES Workshops — These workshops are designed to help patients develop appropriate behaviors to deal with stigmatizing situations. They will focus on three main areas: adapted physical activities, nutrition and mental well-being. They will include sessions on developing self-esteem, improving body image and managing emotions. The aim will be to deconstruct the myths and stereotypes surrounding obesity.
  Arms: STEREOBES
Behavioral: Un Poids en moins — Standard intervention proposed by "La Vie la Santé"
  Arms: CONTROL

SUMMARY:
This project proposes to integrate a psychosocial approach into the therapeutic patient education program (TPE) at "La Vie la Santé", an innovative health promotion platform at Poitiers University Hospital. A randomized study will be set up within the active file of patients referred by the specialized obesity center of Poitou-Charentes and integrated into this patient education program (TPE) program. Patients randomized to the TPE-STEREOBES experimental cohort arm will participate for 12 months in obesity-specific adapted physical activity workshops, on the one hand, and in workshops based on "social well-being" on the other, designed as part of this study. They will be assessed when they enter the program (T0), then at 3 months (T3), 6 months (T6), 12 months (T12) and finally 6 months later (T18). Assessments at T0, T12 and T18 will be compared with those of patients in the control group, made up of patients followed up at the specialized obesity center who were not included in the TPE-STEREOBES program.

DETAILED DESCRIPTION:
Obesity is a major public health issue, affecting 17% of the population. It is also a major societal issue, due to the "grossophobia" and discriminatory attitudes to which obese people are subjected. Widely documented in the literature, the "stereotype threat" effect of obesity has negative psychological consequences (e.g. stress, anxiety, reduced self-esteem, deterioration of self-image, impaired cognitive functions), can lead to the adoption of pathogenic behaviors (e.g. energy-dense foods, limitation of physical activity, avoidance of social situations) and therefore generates a deterioration in quality of life. To date, while the psychotherapeutic support of obese patients and the provision of adapted physical activities have been well documented, no intervention targeting the deleterious effects of this obesity stereotype threat has been tested in the medical follow-up of obese patients.

This innovative project aims to develop, implement and evaluate psychosocial interventions to remediate the effects of obesity stereotypes on severely obese patients. Its aim is to improve their sense of self-efficacy, a factor recognized as an antecedent of behavioral and attitudinal changes that contribute to improving their quality of social life and health status. To this end, this project proposes to integrate a psychosocial approach into the therapeutic patient education (TPE) program at "Vie la Santé", an innovative health promotion platform at Poitiers University Hospital. A randomized study will be set up within the active file of patients referred by the Poitou-Charentes specialized obesity center and integrated into this therapeutic patient education (TPE) program. Patients randomized to the ETP-STEREOBES experimental cohort arm will participate for 12 months in obesity-specific APA workshops, on the one hand, and in workshops based on "social well-being" on the other, designed as part of this study. They will be assessed when they enter the program (T0), then at 3 months (T3), 6 months (T6), 12 months (T12) and finally 6 months later (T18). Assessments at T0, T12 and T18 will be compared with those of patients in the control group, made up of patients attending a specialized obesity center who are not included in the ETP-STEREOBES program.

The benefits of this study will be not only individual, but also collective and institutional, by providing the partners and beneficiaries of this research with operational and innovative knowledge, tools and practices contributing to the fight against discrimination, notably via a showcase website and the scientific dissemination of research findings.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30
* Patient affiliated to or benefiting from a social security scheme.

Exclusion Criteria:

* Patient suffering from an uncontrolled psychiatric illness with no suitable treatment in place (e.g. schizophrenia, bipolar disorder, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Obesity-specific personal efficacy | At Baseline, 3 months follow up, 6 months follow up, 12 months follow up, 6 months after the end of the program
  Obesity-specific personal efficacy is recognized in the literature as one of the determinants of attitudinal and behavioral change. This is a 40-item scale grouping together 4 dimensions: Eating Behavior Management (EBM), Physical Activity (PA), Self-Image and How Others See You (SIRA), Social Relations (SR). For each item, the patient indicates a score from 1 "not at all capable" to 10 "completely capable".

SECONDARY OUTCOMES:
Brief Coping Responses Inventory (BCRI-10) | At Baseline, 3 months follow up, 6 months follow up, 12 months follow up, 6 months after the end of the program
  This scale comprises 10 items grouping together 2 dimensions: reappraisal coping and disengagement coping. Items are measured on a scale from 0 (Never) to 4 (Always).
Weight Bias Internalization Scale | At Baseline, 3 months follow up, 6 months follow up, 12 months follow up, 6 months after the end of the program
  Patients indicate on 10 items their degree of agreement with the proposed statements on a 7-point Likert scale ranging from 1 "completely disagree" to 7 "completely agree".
Body Shape Questionnaire (BSQ-14) | At Baseline, 3 months follow up, 6 months follow up, 12 months follow up, 6 months after the end of the program
  This scale measures preoccupation and dissatisfaction with one's body because of weight. It consists of 14 items ranging from 1 (never) to 6 (always).

CONTACTS AND LOCATIONS:
Locations (1):
- Poitiers University Hospital, Poitiers, Vienne, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ramsamy G, Esnard C; STEREOBES Consortium; Mosbah H, Soussi Berjonval D, Faure JP, Albouy M. Effect of a patient education program focused on weight stigma on quality of life and self-efficacy in patients living with obesity: study protocol for a randomized controlled trial. BMC Psychol. 2024 Dec 18;12(1):734. doi: 10.1186/s40359-024-02274-8. PMID 39696393